CLINICAL TRIAL: NCT00008450
Title: Induction of Mixed Hematopoietic Chimerism in Patients With Severe Combined Immunodeficiency Disorders Using Allogeneic Bone Marrow and Post-Transplant Immunosuppression With Cyclosporine and Mycophenolate Mofetil
Brief Title: Total-Body Irradiation Followed By Cyclosporine and Mycophenolate Mofetil in Treating Patients With Severe Combined Immunodeficiency Undergoing Donor Bone Marrow Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1227.00; NCI-2010-02045 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1227.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01HL036444 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2001-01-06; First posted 2001-01-08 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Adenosine Deaminase Deficiency; Autosomal Recessive Disorder; Immune System Disorder; Purine-Nucleoside Phosphorylase Deficiency; Severe Combined Immunodeficiency; Severe Combined Immunodeficiency With Absence of T and B Cells; X-Linked Severe Combined Immunodeficiency
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency; Immune System Diseases; Purine Nucleoside Phosphorylase Deficiency; Severe Combined Immunodeficiency; X-Linked Combined Immunodeficiency Diseases | interventions — Cyclosporine; Cyclosporins; Mycophenolic Acid; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cyclosporine, mycophenolate mofetil, transplant) (Experimental): Patients receive cyclosporine PO or IV on days -3 to 100 followed by a taper until day 180 and mycophenolate mofetil PO or IV on days 0-40 with a taper until day 96 in the absence of unacceptable toxicity. Unrelated donor recipients also undergo TBI on day 0. Patients undergo bone marrow transplant on day 0.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Drug: Cyclosporine; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Undergo allogeneic bone marrow transplant
  Other Names: Allo BMT; Allogeneic BMT
Drug: Cyclosporine — Given PO or IV
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO or IV
  Other Names: Cellcept; MMF
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo nonmyeloablative allogeneic hematopoietic stem cell transplant
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation

SUMMARY:
This pilot clinical trial studies total-body irradiation followed by cyclosporine and mycophenolate mofetil in treating patients with severe combined immunodeficiency (SCID) undergoing donor bone marrow transplant. Giving total-body irradiation (TBI) before a donor bone marrow transplant using stem cells that closely match the patient's stem cells, helps stop the growth of abnormal cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may mix with the patient's immune cells and help destroy any remaining abnormal cells. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To safely establish partial lymphoid chimerism (1-95% donor cluster of differentiation [CD]3+ cells) using a non-lethal conditioning regimen in patients with severe combined immunodeficiency syndrome.

II. To define the kinetics of immune reconstitution following a non-lethal conditioning regimen in patients with immunodeficiency diseases.

OUTLINE:

Patients receive cyclosporine orally (PO) or intravenously (IV) on days -3 to 100 followed by a taper until day 180 and mycophenolate mofetil PO or IV on days 0-40 with a taper until day 96 in the absence of unacceptable toxicity. Unrelated donor recipients also undergo TBI on day 0. Patients undergo bone marrow transplant on day 0.

After completion of study treatment, patients are followed up at 6 months and then yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe combined immunodeficiency syndrome:

  * SCID with presence of B lymphocytes

    * X-linked SCID (presence of B lymphocytes)
    * Autosomal recessive SCID
* Patients with severe combined immunodeficiency syndrome:

  * SCID with absence of T and B lymphocytes
* Patients with severe combined immunodeficiency syndrome:

  * Purine metabolite deficiencies, deficiencies of the purine metabolites

    * Adenosine deaminase (ADA) deficiency
    * Purine nucleoside phosphorylase (PNP) deficiency
* DONOR: Related donor who is human leukocyte antigen (HLA) genotypically identical at least at one haplotype and may be genotypically or phenotypically identical for serological typing for HLA-A, B, C, and at the allele level for DRB1 and DQB1; related donors other than siblings must be matched at HLA-A, B, and C (at highest resolution available at the time of donor selection) and at DRB1 and DQB1 by deoxyribonucleic acid (DNA) typing; if more than one HLA-identical sibling is available, priority will be given to the oldest normal donor
* DONOR: Unrelated donors who are prospectively matched for HLA-A, B, C, DRB1 and DQB1 by DNA typing at the highest resolution routinely available at the time of donor selection; only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing

Exclusion Criteria:

* Patients with viral associated T cell immunodeficiency disorders, such as human immunodeficiency virus (HIV)
* Patients with other disease or organ dysfunction that would limit survival to less than 30 days
* DONOR: Identical twin
* DONOR: Pregnancy
* DONOR: HIV seropositive
* DONOR: A positive anti-donor cytotoxic cross match is absolute donor exclusion
* DONOR: Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-HLA allele mismatch, i.e., the patient is A*0201, and this type of mismatch is not allowed
* DONOR: < 6 months old, > 75 years old

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1997-08-11 (Actual); Primary Completion 2011-10-25 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Mixed hematopoietic chimerism in a population of pediatric patients with immunodeficiency diseases | Up to 5 years
  It will be established whether a non-lethal conditioning regimen can successfully induce mixed hematopoietic chimerism in a population of pediatric patients with immunodeficiency diseases, without adverse effects on mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Burroughs, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States